CLINICAL TRIAL: NCT03444467
Title: A Randomised, Double-blinded, Single Subcutaneous Dose Escalation Trial Investigating the Safety and Tolerability of NNC9204-1513 in Healthy Subjects
Brief Title: First Research Study to Compare a Possible New Medicine NNC9204-1513 to the Medicine Glucagon, in Healthy People.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9513-4290; U1111-1180-8217 (Other: World Health Organization (WHO)); 2016-001173-33 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-02-05; First posted 2018-02-23 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Glucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NNC9204-1513 (Experimental): Participants will receive increasing doses of NNC9204-1513.
  Interventions: Drug: NNC9204-1513; Drug: Placebo
- Glucagon (Active Comparator): Participants will receive a single fixed dose of glucagon.
  Interventions: Drug: Glucagon; Drug: Placebo

INTERVENTIONS:
Drug: NNC9204-1513 — Participants will receive NNC9204-1513 subcutaneous (s.c., in to a skin fold on the stomach) injection as single increasing doses of 0.01 mg, 0.04 mg, 0.10 mg, 0.25 mg, 0.50 mg, 1.0 mg or 2.0 mg. Each participant will only be given one dose.
  Dose escalation will proceed to the next planned dose level if there are no safety concerns raised by the investigator or by the trial safety group.
  Arms: NNC9204-1513
Drug: Glucagon — Participants will receive single dose of 1 mg glucagon s.c. injection.
  Other Names: GlucaGen®
  Arms: Glucagon
Drug: Placebo — Participants will receive single dose of placebo (for double dummy injections).

SUMMARY:
The study is comparing the new medicine NNC9204-1513 with a standard therapy of glucagon (GlucaGen®). This is the first time NNC9204-1513 is given to humans.

Participants will either receive NNC9204-1513 or GlucaGen® - which treatment you get is decided by chance (like flipping a coin). Neither the participant nor the study doctor will know which study medicine (NNC9204-1513 or GlucaGen®) the participant is receiving (double -blinding). In case of emergency, this information will be readily available.

NNC9204-1513 is a new medicine for rescue treatment of severe low blood sugar and currently not available on the market (doctors cannot prescribe this medicine). The participant will receive two or three single injections below the skin. One injection will contain NNC9204-1513 or GlucaGen®. The other injection will include placebo - this is a product that looks like the actual study drug but without any active ingredients. If a third injection is given, this will contain NNC9204-1513 or placebo. NNC9204-1513 and GlucaGen® will be given using different devices and volumes. In order to mask these external differences, a "double dummy" approach will be used, that means when you get either of the study medicine (NNC9204-1513 or GlucaGen®) you will get another injection which contains no medicine called 'placebo' (it will not have any effect on the body). Dependent on the injection volume to be administered, injections are given by either syringe with needle or an injection pen (NovoPen Echo®). The study will last for up to 39 days.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 -55 years (both inclusive), at the time of signing informed consent
* Body mass index (BMI) between 18.5 and 28.0 kg/sqm (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, ECG and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol
* Smoker (defined as a subject who is smoking at least one cigarette or equivalent daily) who is not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period
* Any blood draw in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | from time of dosing (day 1) to completion of the safety follow-up visit (day 8)
  Count of events

SECONDARY OUTCOMES:
Change from baseline in haematology | baseline (day 1), follow-up visit (day 8)
Change from baseline in biochemistry | baseline (day 1), follow-up visit (day 8)
Change from baseline in fibrinogen | baseline (day 1), follow-up visit (day 8)
  measured in g/L
Change from baseline in lipids | baseline (day 1), follow-up visit (day 8)
Change from baseline in glucose metabolism | baseline (day 1), follow-up visit (day 8)
Change from baseline in hormones | baseline (day 1), follow-up visit (day 8)
Change from baseline in urine dipstick parameter | baseline (day 1), follow-up visit (day 8)
Change from baseline in systolic- and diastolic blood pressure | baseline (day 1), follow-up visit (day 8)
  Measured in mm Hg
Change from baseline in body temperature | baseline (day 1), follow-up visit (day 8)
Change from baseline in respiration rate | baseline (day 1), follow-up visit (day 8)
Change from baseline in 12-lead electrocardiogram (ECG) heart rate | baseline (day 1), follow-up visit (day 8)
Change from baseline in 12-lead ECG (RR interval) | baseline (day 1), follow-up visit (day 8)
Change from baseline in 12-lead ECG (PR interval) | baseline (day 1), follow-up visit (day 8)
Change from baseline in 12-lead ECG (QRS interval) | baseline (day 1), follow-up visit (day 8)
Change from baseline in 12-lead ECG (QT interval) | baseline (day 1), follow-up visit (day 8)
Change from baseline in 12-lead ECG (QTc intervals [Fridericia]) | baseline (day 1), follow-up visit (day 8)
  QT interval corrected for heart rate by Fridericia's formula
Change from baseline in Physical examination | baseline (day 1), follow-up visit (day 8)
Incidence of injection site reactions | After administration of the trial products (day 1) until completion of the post-treatment follow-up visit (day 8).
AUC0-15min,SD, area under the plasma concentration time curve | 0 to 15 minutes after single dose
t1/2,SD, terminal half-life | Measured for 24 hours after administration of a single s.c. dose
Onset of appearance | Measured for 24 hours after administration of a single s.c. dose
  Time from trial product administration until first time plasma concentration ≥ lower limit of quantification (LLOQ)
AUCPG,0-15min,SD, area under the plasma glucose time curve | 0 to 15 minutes after single dose
ΔPG0-15min,SD, Increase in plasma glucose concentration from 0 to 15 minutes | 0 to 15 minutes after single dose
  Calculated as: Plasma glucose concentration at 15 minutes after single dose minus plasma glucose concentration at 0 minute
Change from baseline in 12-lead ECG (overall evaluation) | baseline (day 1), follow-up visit (day 8)
Change from baseline in prothrombin time | baseline (day 1), follow-up visit (day 8)
  measured in seconds
Change from baseline in Activated Partial Thromboplastin time (APTT) | baseline (day 1), follow-up visit (day 8)
  measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://www.novonordisk-trials.com/